CLINICAL TRIAL: NCT00281125
Title: A Two-Cohort Phase I/II Trial of PTK787 and Pemetrexed With or Without Cisplatin in Patients With Advanced Non-Small Cell Lung Cancers and Malignant Pleural Mesotheliomas
Brief Title: Phase I/II Trial of PTK787 and Pemetrexed With or Without Cisplatin for Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Suspended due to data issues revealed at DSMB meeting. Planned amendment but was never submitted. Study was then closed.
Sponsor: Nevada Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NVCI05-14
Record Dates: First submitted 2006-01-06; First posted 2006-01-24 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Non-Small Cell Lung Cancer and Pleural Mesothelioma
Keywords: Non-Small Cell Lung Cancer; Pleural Mesothelioma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Mesothelioma, Malignant | interventions — vatalanib; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: PTK787 and Pemetrexed with or without Cisplatin

SUMMARY:
This is an open-label, two-arm, multicenter Phase IA/II dose-escalation study of PTK787 in combination with Pemetrexed alone (Cohort 1) or Pemetrexed and Cisplatin (Cohort 2).

This study is designed to determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of PTK787 when administered in combination with Pemetrexed or Pemetrexed and Cisplatin, and to characterize the safety, tolerability, biologic activity, and PK profile of PTK787 in adult patients with advanced non-small cell lung cancers and mesotheliomas.

DETAILED DESCRIPTION:
This is an open-label, two-arm, multicenter Phase IA/II dose-escalation study of PTK787 in combination with Pemetrexed alone (Cohort 1) or Pemetrexed and Cisplatin (Cohort 2).

This study is designed to determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of PTK787 when administered in combination with Pemetrexed or Pemetrexed and Cisplatin, and to characterize the safety, tolerability, biologic activity, and PK profile of PTK787 in adult patients with advanced non-small cell lung cancers and mesotheliomas.

In cohort 1, PTK787 will be administered orally every 12 hours on days 2-42 of a 42-day cycle. In addition, Pemetrexed will be administered on days 1 and 22.

In cohort 2, PTK787 will be administered orally every 12 hours on days 2-42 of a 42 day cycle. In addition, Pemetrexed will be administered on days 1 and 22. Thirty minutes after Pemetrexed administration, Cisplatin will be infused on days 1 and 22.

In the current study, initially patients will be treated on Cohort 1 (Pemetrexed + PTK787). Once an MTD determination is made on this cohort (or PTK787 has been escalated to the maximum dose of 750 mg Q12h enrollment will begin on Cohort 2. At the MTD dose, both cohorts will be expanded to a minimum of 20 patients to determine additional safety of the combinations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced non-small cell lung cancers (non-squamous variety and advanced mesotheliomas
* Patients with advanced solid tumors who are refractory to standard treatments and/or standard treatments are not be available for the patient

Exclusion Criteria:

* Non-small cell carcinoma of squamous variety
* Patients with uncontrolled brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-01; Primary Completion 2006-09 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To determine the Maximum tolerated dose (MTD) and Dose Limiting toxicities (DLTs) of a combination of Pemetrexed and PTK787/ZK222584 (Cohort 1) and a combination of Pemetrexed with Cisplatin and PTK787/ZK222584 (Cohort 2) in patients

SECONDARY OUTCOMES:
To determine the preliminary evidence of safety of the above combinations in patients with non-small cell lung cancers and/or mesotheliomas (in the expansion cohorts)
To determine the pharmacokinetics of PTK787/ZK222584 in combination with Pemetrexed and Cisplatin
To determine the pharmacokinetics of Pemetrexed in combination with PTK787/ZK 222584
To determine the effect of therapy with the combination on plasma levels of VEGF A, B, C and D and on plasma levels of soluble VEGF-R2.
To determine the relationship between PTK787/ZK 222584 and Pemetrexed pharmacokinetics and plasma levels of VEGF A, B, C, D, soluble VEGF-R2, and exploratory chemotherapeutic response biomarkers.
To determine the baseline expression of VEGF-R2 by immunohistochemistry in patients where paraffin blocks/slides are available.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Sharma, MD, Principal Investigator — Nevada Cancer Institute
Locations (1):
- Nevada Cancer Institute, Las Vegas, Nevada, United States